CLINICAL TRIAL: NCT03352570
Title: Safe (Safe Anastomosis Feasibility Evaluation)-1 Study : a Study to Investigate the Efficacy, Mechanism of Action and Safety of the Colovac Colorectal Anastomosis Protection Device First-In-man Clinical Investigation Study
Brief Title: a Study to Investigate the Efficacy, and Safety of the Colovac Colorectal Anastomosis Protection Device.
Acronym: SAFE-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Safeheal (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: SAFE-1
Record Dates: First submitted 2017-11-13; First posted 2017-11-24 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Gastrointestinal Anastomotic Complication
Keywords: anastomotic leakage; fistula
MeSH Terms: conditions — Anastomotic Leak; Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COLOVAC device (Experimental): colorectal surgery performed per standard of care with deployment of the Colovac device to protect the anastomosis site
  Interventions: Device: COLOVAC

INTERVENTIONS:
Device: COLOVAC — The intervention consists in the placement of the Colovac device, during the colorectal surgery, Once the colorectal anastomosis has been completed as per standard care and the water-thightness of the anastomosis has been verified.

SUMMARY:
The purpose of this study is to evaluate theColovac device, a single use, temporary intraluminal bypass device,intended to reduce contact of fecal content with an anastomotic site, following colorectal surgery (open or laparoscopic).

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be >= 18 and <= 65 years old
2. Indicated for colorectal resection
3. Patient has been assessed by a multi-disciplinary team and it was determined that as per standard of care, they are eligible to bear a diverting ostomy
4. Willing to comply with protocol-specified follow-up evaluations
5. Signed Informed Consent

Exclusion Criteria:

1. Patient with inflammatory bowel disease
2. Pregnant or nursing female subject (a pregnancy test should be conducted the day prior to the procedure for all women in age of procreating)
3. Known allergy to nickel or other components of the Colovac kit
4. Any significant medical condition which, in the investigator's opinion, may interfere with the subject's optimal participation in the study, including:

   1. immunodeficiency
   2. steroid therapy
   3. infections at the time of intervention
   4. major surgical or interventional procedures within 30 days prior to this study or planned surgical or interventional procedures within 30 days of entry into this study
   5. diagnosis of bowel obstruction, bowel strangulation, peritonitis, bowel perforation, local or systemic infection, ischemic bowel, carcinomatosis
   6. preexisting sphincter problems or evidence of extensive local disease in the pelvis
   7. blood loss (> 500 cc)
   8. non amended peroperative anastomosis failure
   9. intra-operative adverse events
   10. malnourishment
   11. obesity (BMI > 35)
   12. history of excessive smoking and alcohol use
5. The subject is currently participating in another investigational drug or device study that has not completed the primary endpoint or that clinically interferes with the endpoints of this study
6. Patient unable to give consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2018-09-26 (Actual); Study Completion 2019-03-26 (Actual)

PRIMARY OUTCOMES:
Rate of adverse events | up to 3 months
  occurence of intraoperative and postoperative complications

SECONDARY OUTCOMES:
device introduction success rate | During surgery
  Ability to introduce, deploy and retrieve the Colovac Anastomosis Protection Device in/from the desired location in the colon
Device placement success rate | During surgery
  Measured by number of successful placement divided by overall placement number
Colovac procedure time | During surgery
  Procedure duration measured in minutes
Migration rate of the Colovac device | During surgical procedure and up to 15 days after placement
  defined by the number of devices migrated over the anastomosis divided by the number of devices placed
Device retrieval success rate | At 14 days after device placement
  Retrieval success rate measured by number of successful retrieval without complication divided by overall number of retrieval performed
rate of digestive disorders | up to 15 days after surgery
  Measured as number of patients presenting digestive disorders divided by overall number of patients
level of patient comfort measured using NIH's PROMIS health measurement questionnaires | up to 15 days after surgery
  measures using health measurement questionnaires to assess parameters like pain (visual analogue scale - 1 : no pain - 10 : worse pain ever); bowel incontinence (visual analogue scale - 1 : no incontinence - 10 : uncontrollable incontinence), diarrhea (visual analogue scale - 1 : no pain - 10 : worse pain ever); bowel incontinence (visual analogue scale - 1 : no diarrhea - 10 : more than 3 episodes of diarrhea per day)
occurence of anastomosis leakage | up to 3 months after initial surgery
  measured as mean number of anastomosis leakage episodes per patient
occurrence of anastomosis fistula | up to 3 months after initial surgery
  measured as mean number of anastomosis fisutal episodes per patient
occurrence of anastomotic abcesses | up to 3 months after initial surgery
  measured as mean number of anastomosis abcess episodes per patient

CONTACTS AND LOCATIONS:
Locations (3):
- UZA Antwerp, Antwerp, Belgium
- France (2):
  - Hopital Saint-Antoine, Paris
  - Ihu Strasbourg, Strasbourg

IPD SHARING:
Plan to Share IPD: Undecided